CLINICAL TRIAL: NCT00638274
Title: Comparison of Loss of Resistance Technique With Air Versus Saline to Identify Epidural Space for Combined Spinal Epidural Labor Analgesia
Brief Title: Comparison of Loss of Resistance Techniques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Air versus Saline
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Pain Relief
Keywords: Quality of pain relief with 2 different methods of identifying epidural space
MeSH Terms: interventions — Air; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Air (Active Comparator): Air 3 ml used to identify epidural space
  Interventions: Procedure: Air
- Saline (Active Comparator): Saline 3 ml used to identify epidural space
  Interventions: Procedure: Saline

INTERVENTIONS:
Procedure: Air — 3 mls used for identifying epidural space
  Arms: Air
Procedure: Saline — 3 mls of saline used to identify epidural space
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether there is a difference in success outcome of the combined spinal epidural labor analgesia between air versus saline when used to identify the epidural space.

DETAILED DESCRIPTION:
When the epidural needle is inserted initially, it is typically connected to a syringe filled with 2-3 ml or air or saline. This is used to help identify the placement of the epidural needle. Both air and saline are commonly used and it is not clear and debatable which is a better method to identify the correct placement of the needle. Some doctors like using air in the syringe because when a drop of clear fluid returned from the smaller spinal needle, it would be clear to indicate the correct space for first dose of medicine since no pre-existing fluid was used. In group Saline, 3 mL of saline will be used. In group Air, 3 mL of air will be used in the syringe during the procedure.

The medicine will be administered in the usual manner the doctor has identified the correct location for administration. The amount of pain during labor will be assessed the patient giving a number from 0 to 10 with 0 being no pain and 10 being the worst pain.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females weighing less than or equal to 250 lbs
* Request for neuraxial labor analgesia

Exclusion Criteria:

* ASA physical status greater than II

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2005-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Pan, MSEE, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-AIR: Air 3 ml used to identify epidural space
  Air: 3 mls used for identifying epidural space
- 2-SALINE: Saline 3 ml used to identify epidural space
  Saline: 3 mls of saline used to identify epidural space
Period: Overall Study
Arm/Group | 1-AIR | 2-SALINE
Started | 179 | 177
Completed | 173 | 172
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-AIR | 2-SALINE | Total
Number analyzed (Participants) | 173 | 172 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 173 | 172 | 345
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 172 | 345
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 173 | 172 | 345

OUTCOME MEASURES:

1. Primary Outcome: Success of Spinal Labor Analgesia From Combined Spinal Epidural
Description: Number of participants that had successful spinal labor analgesia in each group.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1-AIR | 2-SALINE
Number analyzed (Participants) | 173 | 172
Participants | 163 | 161
Statistical Analysis 1: Comparison: 1-AIR; Test type: Other; p > .05, Chi-squared
Statistical Analysis 2: Comparison: 2-SALINE; Test type: Other; p > .05, Chi-squared

2. Secondary Outcome: Number of Participants With Failed Epidural Catheters
Description: Number of Participants with Failed Epidural Catheters and that had to be replaced at any time measured from the time of the catheter is placed until the time of delivery.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1-AIR | 2-SALINE
Number analyzed (Participants) | 173 | 172
Participants | 5 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the epidural catheter was placed until the time of delivery, usually less than 24 hours
Arm/Group | 1-AIR | 2-SALINE
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/172
Other Adverse Events (participants affected / at risk) | 0/173 | 0/172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-10-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT00638274/Prot_SAP_000.pdf